CLINICAL TRIAL: NCT06351813
Title: Predicting Adverse Kidney Events of Cardiac Surgery-Associated Acute Kidney Injury Using Novel Biomarkers--A Multicenter Observational Study
Brief Title: Predicting Adverse Kidney Events of Cardiac Surgery-Associated Acute Kidney Injury Using Novel Biomarkers
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Zhongshan Hospital (Xiamen), Fudan University (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guowei Tu, Professor, Shanghai Zhongshan Hospital
Other Study IDs: B2024-029R
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury; Critical Illness; Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serial blood and urine samples for biomarker analysis were collected after surgery and then every 6 h in day 1 and then daily until discharge from ICU or for a maximum of 7 days, respectively. Plasma (EDTA), serum, and urine supernatants were frozen within 2 h of sample collection, stored at -80℃, and thawed immediately before analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to identify and validate novel biomarkers for predict acute kidney injury (AKI) subphenotype, major adverse kidney events and other poor outcomes.

DETAILED DESCRIPTION:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a serious condition that is associated with increased mortality and morbidity. However, the current criteria for assessing the severity of AKI may not adequately capture the heterogeneity of this condition. This can lead to difficulties in identifying treatment effects in specific patient subgroups, which may contribute to the growing number of negative interventional trials in AKI. To address this issue, researchers have developed and validated two subphenotypes of AKI: resolving and nonresolving. These subphenotypes are based on the trajectory of serum creatinine (SCr) levels in the first 3 days after hospital presentation. By stratifying AKI patients based on these subphenotypes, we can better assess their risk and predict outcomes.

Several novel biomarkers have been developed to aid in the early detection of AKI, discrimination of its underlying causes, and prediction of outcomes. However, it remains unclear whether these biomarkers can accurately predict the development of a nonresolving AKI subphenotype. In our present study, we aim to address this gap in knowledge by conducting a large cohort study. Our goal is to identify and validate novel biomarkers that can effectively detect the resolving subphenotype of AKI, as well as predict major adverse kidney events and other poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery who experienced AKI within 48 hours of cardiac surgery were screened.

Exclusion Criteria:

* History of End Stage Renal Disease or on Dialysis;
* prior kidney transplantation;
* patients with a DNR order;
* patients without written informed consent;
* pregnancy;
* moribund patients with expected death within 24 h or whose survival to 28 days was unlikely due to an uncontrollable comorbidity (i.e., end-stage liver or heart disease, untreatable malignancy)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with age ≥ 18 years who experienced AKI within 48 hours of cardiac surgery were included in this study.
Sampling Method: Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
AKI nonresolving subphenotype | 7 days
  The resolving subphenotype was defined by a decrease of 0.3 mg/dl or 25% in SCr from its maximum during the first 3 days of study enrollment. All subjects with AKI who did not meet this criterion were classified as having a nonresolving subphenotype

SECONDARY OUTCOMES:
Major adverse kidney events at 30 days | 30 days
  Major adverse kidney events (MAKE) was defined as the composite of≥25% loss in estimated glomerular filtration rate (eGFR), dialysis, or death. Estimated GFR was calculated from serum creatinine using the MDRD equation.
Major adverse kidney events at 90 days | 90 days
  MAKE was defined as the composite of≥25% loss in estimated glomerular filtration rate (eGFR), dialysis, or death. Estimated GFR was calculated from serum creatinine using the MDRD equation.
Major adverse kidney events at 365 days | 365 days
  MAKE was defined as the composite of≥25% loss in estimated glomerular filtration rate (eGFR), dialysis, or death. Estimated GFR was calculated from serum creatinine using the modification of diet in renal disease (MDRD) equation.
Mortality | 365 days
  Mortality at 30 days, 90 days and 365 days
Receipt of renal replacement treatment | 365 days
  Patients received renal replacement treatment during hospital stay
Moderate and severe AKI | 7 days
  Kidney Disease Improving Global Outcomes (KDIGO) stage 2 or stage 3
AKI progression | 7 days
  worsening of KDIGO stage within 1 week (progressing from stage 1 to either stage 2 or stage 3, or from stage 2 to stage 3).
  Patients diagnosed with progressive or persisting stage 3 AKI (stage 3 AKI for >3 consecutive days) were classified as having AKI progression.
  If patients who presented with stage 3 AKI but not requiring RRT subsequently required dialysis or developing persist severe AKI or death within 7 days, this was considered progression.
Composite Outcome | 30 days
  Stage 3 AKI, renal replacement therapy or death through outpatient or telephone follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Professor, Study Director — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No